CLINICAL TRIAL: NCT00726583
Title: A Phase I Trial of Oral PX-866 (a PI-3K Inhibitor) in Patients With Advanced Solid Tumors
Brief Title: Phase I Trial of Oral PX-866
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-866-001
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2011-10

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Solid Tumors; Carcinoma; PI-3K; PI3 kinase; PI3K
MeSH Terms: conditions — Neoplasms; Carcinoma; Hereditary Sensory and Autonomic Neuropathies | interventions — PX-866

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Drug (Experimental): Dose Escalation
  Interventions: Drug: PX-866

INTERVENTIONS:
Drug: PX-866 — Oral solution, dose escalation, once per day on days 1 to 5 and 8 to 12 or days 1-28 of a 28 day cycle, until progression or development of unacceptable toxicity

SUMMARY:
This study is being conducted to determine the safety and maximally tolerated dose of PX-866 when given orally on two different schedules: daily on days 1-5 and 8-12 of a 28 day cycle and daily on days 1-28 of a 28 day cycle.

DETAILED DESCRIPTION:
PX-866 is a targeted inhibitor of PI-3K. This study is being conducted to determine the maximally tolerated dose of PX-866 when given orally on two different schedules: daily on days 1-5 and 8-12 of a 28 day cycle and daily on days 1-28 of a 28 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced solid tumor and has failed or is intolerant of standard therapy, or for whom standard therapy does not exist.
* 18 years of age or older.
* ECOG performance status 0 to 1.
* Predicted life expectancy of at least 12 weeks.
* Discontinued prior chemotherapy or other investigational agents for at least three weeks prior to receiving the first dose of study drug (six weeks for mitomycin C, nitrosureas,vaccines,or antibody therapy)and recovered from the toxic effects of the prior treatment (recovered to baseline or ≤grade 1 per Common Toxicity Criteria for Adverse Events (CTCAE)).
* Discontinued any radiation therapy for at least four weeks and have recovered from all radiation-related toxicities (recovered to baseline or ≤CTCAE grade 1) prior to receiving the first dose of study drug. Palliative radiation of 10 fractions or less is permitted and a four week interval is not necessary (also allowed during therapy).
* Adequate hematologic function as defined by the following: WBC count >3,000 cells/μL; platelets >100,000/μL; hemoglobin >9 g/dL (may be transfused to this level); ANC >1500 cells/μL.
* Adequate hepatic function as defined by the following: bilirubin <1.5 mg/dL; aspartate aminotransaminase (AST/SGOT) & alanine aminotransferase (ALT/SGPT) <2.5 x ULN or <5 x ULN if due to metastatic disease.
* Adequate renal function as defined by serum creatinine level <1.5 mg/dL.

Exclusion Criteria:

* Any active infection at study entry.
* Known diabetes or fasting blood glucose>160 mg/dL.
* Known human immunodeficiency virus (HIV).
* Any serious concomitant systemic disorders that in the opinion of the investigator would place the patient at excessive or unacceptable risk of toxicity.
* Surgery within the four weeks prior to the first dose
* Significant central nervous system (CNS) or psychiatric disorder(s) that preclude the ability of the patient to provide informed consent.
* Known or suspected brain metastases that have not received adequate therapy or for which the patient requires treatment with steroids or anticonvulsants. In the case of previously treated brain metastases, a minimum four week interval between completion of radiation therapy and registration on study with radiologic evidence of stable or responding brain metastases is required. In the setting of previous CNS metastasectomy, adequate (minimum four week) recovery from surgery and/or radiation therapy should be documented.
* Leptomeningeal brain metastases should be excluded regardless of whether the metastases have been treated or not.
* History of seizures, non-healing wounds, or arterial thrombosis.
* Unstable atrial or ventricular arrhythmias requiring control by medication; any cardiac ischemic event experienced within the preceding six months; prior history of congestive heart failure requiring therapy.
* Breastfeeding or pregnant (confirmed by serum β-HCG within 10 days prior to the start of study treatment if applicable).
* Total gastrectomy, partial bowel obstruction or any gastrointestinal condition that may interfere with absorption of the study medication.
* Any condition that could jeopardize the safety of the patient and compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Determine the MTD of PX-866 | 28 days
Evaluate the safety profile of PX-866 | 28 days
Evaluate pharmacodynamic measures of the effects of PX-866 on the phosphatidylinositol-3 kinase (PI-3K) pathway and related tumor markers. | 28 days
Determine the PK profile of PX-866. | 28 days

SECONDARY OUTCOMES:
Evaluate the anti-tumor activity of PX-866 in patients with advanced malignancies. | 56 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - M.D. Anderson Cancer Center, Houston, Texas